CLINICAL TRIAL: NCT07081087
Title: Multi-Center Clinical Trial to Replace BM Analysis of Cytopenia by a Peripheral Blood Assay
Brief Title: Replacing Bone Marrow Diagnostics With Peripheral Blood Analysis in MDS/Cytopenia Patients
Status: Recruiting | Type: Observational
Sponsor: Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Other Study IDs: PERIBLODD-MDS
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-09

CONDITIONS: Cytopenia
MeSH Terms: conditions — Cytopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- PERIBLOOD
  Interventions: Diagnostic Test: PERIBLOOD

INTERVENTIONS:
Diagnostic Test: PERIBLOOD — In the study, peripheral blood will be taken from all patients, shipped and analyzed at the Weizmann Institute of Science to produce a report based on our technology. The report will contain data on the diagnosis, blast counts and karyotype. This information will be compared with the results from the bone marrow scan, taken separately to each patient, to validate the accuracy of our technology

SUMMARY:
This study aims to validate a novel, non-invasive diagnostic approach for blood and bone marrow malignancies using single-cell RNA sequencing of circulating hematopoietic stem and progenitor cells (cHSPCs) from peripheral blood. Building on prior work defining normal cHSPC profiles in healthy individuals, the study introduces a pipeline for identifying blood pathologies, with a focus on improving the diagnosis and subclassification of myelodysplastic syndromes (MDS). A multi-center clinical trial is proposed to evaluate the method's ability to predict bone marrow results in patients with cytopenia, potentially reducing reliance on bone marrow biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Platelets < 150 × 109/L or
* Absolute neutrophil count < 1.8 × 109/L or
* Hemoglobin (Hgb) < 13 g/dL (males) and < 12 g/dL (female) and
* For all genders, no evidence of Iron, folinic acid, or B12 deficiency
* All subjects should be referred for BM analysis

Exclusion Criteria:

* Previous diagnosis of leukemia (AML, MPN, ALL, CLL, MGUS/MM or any other gammopathy)
* Lymphocytes>5000/ul
* If patients are recruited after
* Diagnosis of any disease related therapy 3 month prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cytopenia, or suspicion for cytopenia, who are referred to BM from the primary care clinic will be recruited to the study
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of scRNAseq of peripheral blood CD34 cells in the diagnosis of cytopenia | Three months following the peripheral blood sample
  The accuracy of scRNA-seq analysis of peripheral blood CD34-positive cells, together with machine learning algorithms, will be compared with that of bone marrow sampling in cytopenia patients, in order to further validate the reference model that was recently published (https://www.nature.com/articles/s41591-025-03716-5). Among the parameters that will be compared are the diagnosis, blast count, and mutational data

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California San Diego, San Diego, California
  - University of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No